CLINICAL TRIAL: NCT05335031
Title: Ozanimod (Zeposia®) In Patients With RRMS: A 3-Year, Multicenter, Prospective, Non-Interventional Study to Document Utilization, Effectiveness and Quality of Life in Clinical Practice in Germany (OZEAN)
Brief Title: A Study Investigating the Utilization, Effectiveness and Quality of Life in Clinical Practice in Germany for Participants With Relapsing-remitting Multiple Sclerosis Treated With Ozanimod (Zeposia®)
Acronym: OzEAN
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: RPC-1063-MS-003
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis; Relapsing-Remitting; Ozanimod; Zeposia®
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — ozanimod

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Participants with relapsing-remitting multiple sclerosis (RRMS) treated with Ozanimod
  Interventions: Drug: Ozanimod

INTERVENTIONS:
Drug: Ozanimod — As per product label

SUMMARY:
The purpose of this study is to collect real-world data and to gain insights about long-term usage of ozanimod (Zeposia ®), its effect on well-defined outcome parameters comprising participant-relevant outcomes, as well as quality of life, effectiveness, and incidence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of relapsing-remitting multiple sclerosis (RRMS)
* The decision upon treatment with ozanimod must have been made before enrollment and independently of this non-interventional observational study
* All data on ozanimod treatment are collected prospectively. The retrospective documentation of ozanimod therapy and enrollment of participants that are already on ozanimod therapy is not allowed

Exclusion Criteria:

* Special warnings, precautions and contraindications specified in the current version of the Summary of Product Characteristics (SmPC)
* Hypersensitivity to the active substance(s) or to any of the excipients of ozanimod as specified in the prescribing information must not be enrolled
* Participation in any other clinical studies

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 450 relapsing-remitting multiple sclerosis (RRMS) adult participants (any gender) who are either newly treated RRMS participants or who switched from other RRMS treatments to ozanimod are planned to be enrolled in up to 100 specialist study sites (office-based neurologists and clinics) across Germany.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Proportion of participants persistence with therapy | Up to 36 months

SECONDARY OUTCOMES:
Distribution of participant demographics characteristics: Age | At baseline
Distribution of participant demographics characteristics: Sex | At baseline
Distribution of participant demographics characteristics: Height | At baseline
Distribution of participant demographics characteristics: Body weight | At baseline
Distribution of clinical characteristics: Smoking status | At baseline
Distribution of clinical characteristics: Multiple Sclerosis (MS) diagnosis | At baseline
Distribution of clinical characteristics: MS anamnesis/history | At baseline
Distribution of clinical characteristics: Prior diseases | At baseline
Distribution of clinical characteristics: Concomitant diseases | At baseline
Distribution of clinical characteristics: Concomitant medication | At baseline
Distribution of clinical characteristics: Prior MS medication | At baseline
Distribution of clinical characteristics: Physical examination | At baseline
Distribution of clinical characteristics: Reasons for switch to ozanimod | At baseline
Distribution of clinical characteristics: Treatment start with ozanimod | At baseline
Distribution of clinical characteristics: Discontinuation, defined as physician's documentation of a discontinuation of ozanimod treatment | Up to 36 months
Distribution of clinical characteristics: Reason for discontinuation | Up to 36 months
Distribution of clinical characteristics: Subsequent MS treatment | Up to 44 months
Distribution of clinical characteristics: Persistence with therapy | Up to 36 months
Distribution of clinical characteristics: Adherence to therapy | Up to 36 months
Treatment Satisfaction Questionnaire for Medication (TSQM v1.4) | Up to 44 months
Symbol Digit Modalities Test (SDMT) | Up to 44 months
Fatigue scale for motor and cognitive functions (FSMC) | Up to 44 months
Multiple Sclerosis Quality of Life-54 (MSQOL-54) | Up to 44 months
United Kingdom Neurological Disability Rating Scale (UNDS) | Up to 44 months
Clinical Relapse defined as the annualized relapse rate (ARR) | Up to 44 months
Expanded disability status scale (EDSS) | Up to 44 months
Work Productivity and Activity Index-Multiple Sclerosis (WPAI-MS German v2.1) | Up to 44 months
Multiple Sclerosis Health Resource Survey (MS-HRS 3.0) | Up to 44 months
Incidence rate for Adverse Events (AEs) | Up to 44 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Universitätsklinikum Dresden, MS Ambulanz, Dresden, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ziemssen T, Richter S, Maurer M, Buttmann M, Kreusel B, Poehler AM, Lampl M, Linker RA. OzEAN Study to Collect Real-World Evidence of Persistent Use, Effectiveness, and Safety of Ozanimod Over 5 Years in Patients With Relapsing-Remitting Multiple Sclerosis in Germany. Front Neurol. 2022 Jun 27;13:913616. doi: 10.3389/fneur.2022.913616. eCollection 2022. PMID 35832177
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/office-global-policy-and-strategy/fda-recalls-market-withdrawals-safety-information